CLINICAL TRIAL: NCT07097818
Title: Efficacy of Glycemic Improvement Project (GLITTER Study) in Type 1 Diabetes-GLITTER Study 2: a Multicentre, Cluster-randomized, Controlled Trial
Brief Title: Efficacy of Glycemic Improvement Project (GLITTER Study) in Type 1 Diabetes-GLITTER Study 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Xia Li, Professor, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KYZ20250019
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Comprehensive management; T1D teams; Structured education; Peer resources; Diabetes technologies; Glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients with T1D in the intervention group will undergo comprehensive management.
  Interventions: Behavioral: T1D team, structured education, peer support , and diabetes technologies
- Control group (Other): Patients with T1D in the control group will receive routine management.
  Interventions: Behavioral: Routine Management

INTERVENTIONS:
Behavioral: T1D team, structured education, peer support , and diabetes technologies — Patients with T1D will use insulin pumps and CGM , while undergoing structured education courses under the management of a specialized T1D team and engaging in peer support activities.
  Arms: Intervention group
Behavioral: Routine Management — Patients with T1D will be managed according to the routine diagnosis and education model of each hospital.
  Arms: Control group

SUMMARY:
The GLITTER Study 2 is a cluster randomized trial that will evaluate the impact of comprehensive and intensive management, comprising a team, technology, education, and peer resources, on metabolic control and psychological outcomes in patients with type 1 diabetes.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is a lifelong metabolic disease with an increasing disease burden. Despite continuous advancements in diagnostic and treatment technologies, patients of all age groups fail to meet the glycemic targets. Currently, there is a common deficiency in the management of T1D both domestically and internationally, which is specifically manifested as: the disconnection between blood glucose monitoring and insulin adjustment, low utilization rate of new technologies, insufficient patient self-management training, and the absence of psychological intervention, etc.

This GLITTER Study 2 extends the GLITTER Study (Glycemic Improvement with Team, Technology, Education and Peer Resources in type 1 diabetes) by implementing its philosophy (Team, Technology, Education, Peer Resources) to develop a comprehensive T1D management model, integrating these components to enhance management and evaluate effectiveness.

This multicentre, cluster-randomized controlled trial will be conducted across 10 hospitals. It aims to enroll patients with T1D aged ≥6 years who have had the disease for >3 months. Five hospitals were randomly assigned to the comprehensive management intervention group, and five to the usual care group. A total of 400 individuals were recruited into the study. The intervention for the intervention group includes: T1D team (dedicated T1D physicians, certified diabetes educators, registered dietitians), centralized structured education (courses, short videos, and structured educational materials), peer support (volunteer matching, camp, volunteer peer live streaming), and diabetes technologies (insulin pumps and continuous glucose monitoring). The control group received usual care, with the five assigned hospitals continuing their clinical practice. This 52-week trial includes assessments at the following timepoints: screening, week 13 (visit 2), week 26 (visit 3), week 39 (visit 4), and week 52 (visit 5). Throughout the study period, we will evaluate the model's impact on glycemic control and psychosocial outcomes, aiming to establish an evidence-based clinical practice paradigm for T1D management.

ELIGIBILITY:
Eligibility criteria for study hospitals:

1. Members of the China Diabetes Type 1 Study (CD1S).
2. Experience in type 1 diabetes management: treat more than 50 T1D patients per year and have held camp activities at least once.
3. Have type 1 diabetes educators.

Eligibility criteria of study participants:

1. Diagnosis of Type 1 Diabetes.
2. Age ≥6 years, regardless of gender.
3. Duration of disease >3 months.
4. Planned to attend follow-up visits at this hospital within the next year.
5. Possess sufficient cognitive ability to operate all study-related devices.
6. Willing to use continuous glucose monitoring and insulin pumps, upload data, and participate in remote monitoring.
7. Willing to attend structured education sessions and camp activities on time (for the intervention group only).
8. Willing and able to adhere to the study protocol.
9. Willing to sign the informed consent form.

Exclusion Criteria of study participants:

1. Patients who plan to receive diabetes treatment at other hospitals.
2. Patients who have used an automated insulin delivery system or sensor-augmented pump within 3 months prior to screening.
3. Patients who refuse to use continuous glucose monitoring or insulin pumps, or refuse data upload and remote monitoring.
4. Patients with severe cardiovascular, cerebrovascular, hepatic, or renal diseases; uncontrolled systemic diseases, thyroid diseases; autoimmune diseases; or malignancies.
5. Patients diagnosed with hematologic or bleeding disorders.
6. Patients who have received red blood cell transfusions or erythropoiesis-stimulating agents within 3 months prior to screening.
7. Patients who have used any oral, injectable, or intravenous corticosteroids within 8 weeks prior to screening, or who plan to use corticosteroids during the trial.
8. Patients with severe skin diseases that may affect the application sites of continuous glucose monitoring or insulin pump patches.
9. Patients with auditory or visual impairments.
10. Patients with alcohol or drug abuse.
11. Patients who plan to receive blood transfusions during the study period.
12. Patients who plan to undergo elective surgery requiring general anesthesia or dialysis during the study period.
13. Pregnant women, women planning to become pregnant within 1 year of the study, or women who are breastfeeding.
14. Patients who are currently participating in or have participated in other drug or device trials within the last 2 weeks.
15. Patients who, in the investigator's opinion, are not suitable for participation in this clinical trial, such as those with a history of vision impairment, eating disorders, celiac disease, etc.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Baseline, 13, 26, and 52 weeks
  The primary outcome is the Change in Glycated Hemoglobin A1C (HbA1c) before and after the 52 weeks intervention. HbA1c is a physiological marker of the percentage of red blood cells that have glycated (bonded with a sugar). HbA1c is used to measure changes in average blood sugar over the past three months.

SECONDARY OUTCOMES:
Percentage of patients in each group with HbA1c <7.0% | 52 weeks
  HbA1c serves as a crucial physiological marker for assessing average blood sugar levels over the preceding three months. Values below 7.0 are deemed optimal for long-term health. Consequently, a higher number or percentage of individuals achieving an HbA1c level below 7.0 is indicative of a positive outcome, reflecting better glycemic control and reduced risk of complications.
Percentage of patients in each group with HbA1c <7.5% | 52 weeks
  HbA1c serves as a crucial physiological marker for assessing average blood sugar levels over the preceding three months. Values below 7.5 are deemed optimal for long-term health. Consequently, a higher number or percentage of individuals achieving an HbA1c level below 7.5 is indicative of a positive outcome, reflecting better glycemic control and reduced risk of complications.
CGM-measured Percentage Time 70-180 mg/dL (3.9-10.0 mmol/L) | Baseline, 13, 26, and 52 weeks
  The CGM-measured percentage time 70-180 mg/dL (3.9-10.0 mmol/L) refers to the proportion of time during which an individual's blood glucose levels, as continuously monitored by a CGM device. This metric is crucial for assessing glycemic control in individuals with diabetes. Maintaining blood glucose within this target range is associated with better health outcomes and reduced risk of complications.
CGM-measured Percentage Time >180 mg/dL (>10.0 mmol/L) | Baseline, 13, 26, and 52 weeks
  Smaller percentages of CGM-measured time above 180 mg/dL is considered a positive outcome.
CGM-measured Percentage Time >250 mg/dL (>13.9 mmol/L) | Baseline, 13, 26, and 52 weeks
  CGM measured blood sugar values above 250 mg/dL are considered to be undesirable. Thus, less time spent above 250mg/dL is considered a positive outcome.
CGM-Measured Percentage Time <70 mg/dL (<3.9 mmol/L) | Baseline, 13, 26, and 52 weeks
  Blood sugar values measured by CGM that fall below 70 mg/dL are considered potentially hazardous, as they may lead to unconsciousness and, in severe cases, even death. Therefore, minimizing the time spent below 70 mg/dL is regarded as a highly positive outcome, reflecting better management of low blood sugar episodes and enhanced safety for the individual.
CGM-Measured Percentage Time <60 mg/dL (<3.3 mmol/L) | Baseline, 13, 26, and 52 weeks
  Blood sugar values measured by CGM that fall below 60 mg/dL are considered potentially hazardous, as they may lead to unconsciousness and, in severe cases, even death. Therefore, minimizing the time spent below 60 mg/dL is regarded as a highly positive outcome, reflecting better management of low blood sugar episodes and enhanced safety for the individual.
CGM-measured Glucose Standard Deviation (SD) | Baseline, 13, 26, and 52 weeks
  Standard Deviation represents how much glucose levels fluctuate over time from a given average.
CGM-Measured Glucose Coefficient of Variation | Baseline, 13, 26, and 52 weeks
  The Coefficient of Variability (CV) is calculated as the ratio of the standard deviation to the mean of blood sugar values for each participant, as measured by CGM. The reported CV value is derived by multiplying the ratio of the standard deviation to the mean by 100, providing a percentage that reflects the degree of variability in blood sugar levels across the population. A higher CV value, which can range up to 100, signifies greater dispersion of CGM values, indicating more significant fluctuations in blood sugar levels. This increased variability is generally considered an unfavorable outcome, as it may suggest less stable glucose control. Conversely, the minimum CV value is 0, which would indicate no variability in blood sugar levels, representing perfect stability.
CGM-Measured Glucose Risk Index (GRI) | Baseline, 13, 26, and 52 weeks
  The CGM-Measured Glucose Risk Index (GRI) is a comprehensive metric derived from CGM data, designed to quantify the overall risk associated with blood glucose variability. It integrates multiple aspects of glucose levels, including the frequency and severity of both hypo- and hyperglycemic events, as well as the duration of time spent outside the target glucose range. A lower GRI score indicates better glucose stability and lower risk of adverse outcomes related to blood sugar fluctuations.
Self-Management of Type 1 Diabetes for Chinese Adults | Baseline and 52 weeks
  The Self-Management of Type 1 Diabetes for Chinese Adults (SMOD-CA) scale is a validated instrument specifically designed to assess the self-management behaviors and capabilities of adults with type 1 diabetes in the Chinese population. The SMOD-CA consists of 30 items. Responses are rated on a five-point scale, with higher scores indicating better self-management ability. The total score ranges from 0 to 120.
23-item Chinese Version of Self-Report Measure of Self-Management of Type 1 Diabetes for Adolescents | Baseline and 52 weeks
  The 23-item Chinese Version of Self-Report Measure of Self-Management of Type 1 Diabetes for Adolescents (C-SMOD-A-23) is a validated and simplified instrument designed to assess the self-management behaviors and capabilities of adolescents with type 1 diabetes.
Assessment of sleep quality: Pittsburgh Sleep Quality Index | Baseline and 52 weeks
  Pittsburgh Sleep Quality Index (PSQI), a self-report questionnaire comprising seven component scores (subjective sleep quality, sleep latency, duration of sleep, sleep efficiency habits, sleep disturbances, use of sleeping medication, and daytime dysfunction), is used to evaluate sleep quality over the last month.
Hypoglycemic Fear Scale | Baseline and 52 weeks
  The Hypoglycemic Fear Scale is a widely used and validated assessment tool designed to measure the level of fear and anxiety that individuals with diabetes, particularly those with type 1 diabetes, experience in relation to hypoglycemia (low blood sugar).
Diabetes Technology Attitude Scale | Baseline and 52 weeks
  The Diabetes Technology Attitude Scale is a specialized assessment tool designed to evaluate individuals' attitudes toward diabetes-related technologies.
  Tool lists statement and participants reports how much they agree with the statement.
Barriers to Technology | Baseline and 52 weeks
  The Barriers to Technology Questionnaire typically consists of several key sections, each designed to capture different aspects of technology adoption and use.
Diabetes Treatment Satisfaction Questionnaire | Baseline and 52 weeks
  The Diabetes Treatment Satisfaction Questionnaire (DTSQ) is a comprehensive and widely utilized tool designed to assess the level of satisfaction that individuals with diabetes have with their current treatment regimens. The DTSQ is usually administered as a self-report questionnaire, allowing patients to rate their responses on a Likert scale, typically ranging from "very dissatisfied" to "very satisfied." The total score is calculated by summing the responses to all relevant items, with higher scores indicating greater satisfaction with the treatment.
Diagnosis and measurement of the severity of depression: Patient Health Questionnaire | Baseline and 52 weeks
  The Patient Health Questionnaire (PHQ-9) will be used to assess depressive symptoms, including suicidal ideation, over the last two weeks (9 questions). Items are scored 0-3, resulting in a total score of 0-27. Higher scores indicate more symptoms of depression.
Depression Self-Rating Scale for Children | Baseline and 52 weeks
  The Depression Self-Rating Scale for Children (DSRSC) is a standardized psychological assessment tool designed to measure depressive symptoms in children and adolescents. This self-report inventory allows young individuals to rate the frequency and severity of various depressive feelings and behaviors they may be experiencing.
Generalized Anxiety Disorder 7-item scale | Baseline and 52 weeks
  The Generalized Anxiety Disorder 7-item scale (GAD-7) consists of seven items. Each item asks respondents to rate how often they have been bothered by specific anxiety-related symptoms over the past two weeks.
WHO-5 Well-Being Index | Baseline and 52 weeks
  The WHO-5 Well-Being Index (WHO-5) is a brief, self-report questionnaire designed to assess subjective well-being. The WHO-5 consists of five simple and straightforward items. Each item is rated on a 6-point Likert scale, ranging from 0 (not present) to 5 (constantly present). The total score is calculated by summing the responses to all five items, resulting in a score that ranges from 0 to 25. Higher scores indicate better well-being.
Evaluation of the perception of hypoglycemia in the population tested with Clarke score | Baseline and 52 weeks
  Clarke Hypoglycemia Awareness Scores (0-7 score with higher scores associated with impaired awareness).
Evaluation of the perception of hypoglycemia in the population tested with Gold score | Baseline and 52 weeks
  The Gold method is used to assess impaired awareness of hypoglycemia. The scale is from 1 to 7. A score of 4 or more indicates impaired awareness of hypoglycemia.

OTHER OUTCOMES:
Severe hypoglycemic episodes | 52 weeks intervention period
  Frequency of severe hypoglycemic episodes
Diabetes ketoacidosis | 52 weeks intervention period
  Frequency of diabetes ketoacidosis
Serious Adverse Events | 52 weeks intervention period
  Number, nature and severity of serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xia Li, MD, PhD, Principal Investigator — Second Xiangya Hospital of Central South University
Locations (10):
- China (10):
  - Department of Endocrinology and Metabolism, Peking University People's Hospital, Beijing, Beijing Municipality
  - Department of Endocrinology, Quanzhou First Hospital Affiliated to Fujian Medical University, Quanzhou, Fujian
  - Department of Endocrinology, Shenzhen Second People's Hospital, The First Affiliated Hospital of Shenzhen University, Shenzhen, Guangdong
  - Second Department of Endocrinology and Metabolism, Tangshan Gongren Hospital, Tangshan, Hebei
  - Endocrinology and Metabolism Center, The First Affiliated Hospital, and College of Clinical Medicine of Henan University of Science and Technology, Luoyang, Henan
  - Department of Endocrinology, Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Institute of Metabolism and Endocrinology, Second Xiangya Hospital of Centra South University, Changsha, Hunan
  - Department of Endocrinology and Metabolism, Institute of Endocrinology, The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Department of Endocrinology and Metabolism, Laboratory of Diabetes and metabolism research, West China Hospital, Sichuan University, Chengdu, Sichuan
  - Department of Endocrinology, Children's Hospital of Zhejiang University School of Medicine, National Clinical Research Center for Child Health, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No